CLINICAL TRIAL: NCT07244406
Title: A Phase II, Open-Label, Multicenter Clinical Study to Evaluate the Efficacy and Safety of Senl_B19 Autologous Anti-CD19 CAR-T Cells in Subjects With Relapsed or Refractory CD19-Positive B-Cell Acute Lymphoblastic Leukemia
Brief Title: Assessment of Senl_B19 CAR-T Cells in Relapsed/Refractory CD19+ B-ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S1904-201
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: B-ALL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- S1904 CD19 CAR-T (Experimental): Autologous CD19-targeting CAR T cells, dosage 1*10^6/kg, intravenous injection once
  Interventions: Biological: S1904 CD19 CAR-T

INTERVENTIONS:
Biological: S1904 CD19 CAR-T — Autologous CD19-targeting CAR T cells

SUMMARY:
To evaluate the efficacy and safety of S1904 in patients with relapsed or refractory CD19+B-ALL.

DETAILED DESCRIPTION:
The primary objective： To evaluate the efficacy of S1904 in pediatric and adult subjects with relapsed or refractory CD19-positive B-cell acute lymphoblastic leukemia.

The secondary objectives： To further characterize the efficacy and safety profiles of S1904 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* 1.Sign the informed consent and be willing and able to comply with the visit, treatment regimen, laboratory examination and other requirements of the study as stipulated in the trial flow chart; 2.Male or female subjects. Age between 3 and 25 years (inclusive) at the time of ICF signing； 3.Confirmed diagnosis of relapsed/refractory B-ALL at ICF signing; 4.>5% blasts on screening bone marrow biopsy/aspirate; 5.CD19+ malignant cells by flow cytometry (bone marrow or peripheral blood) at screening; 6.Patients with Ph+ ALL are eligible if they meet the relapsed/refractory criteria and have either: failed ≥2 TKI regimens (unless they have a T315I mutation), demonstrated TKI intolerance, or have a contraindication to TKIs; 7.Estimated survival time>3 months.

Exclusion Criteria:

* 1.Relapse of isolated extramedullary disease; 2.Burkitt lymphoma/leukemia； 3.Active acute or moderate-to-severe chronic GVHD within 4 weeks prior to ICF signing. Or, any systemic GVHD treatment within 4 weeks prior to infusion; 4.No uncontrolled active infection at the time of ICF signing or apheresis.; 5.Prior receipt of any CAR-T therapy or other cellular/gene therapy before screening; 6.Received investigational drugs or systemic anti-tumor therapy within 4 weeks or 5 half-lives (whichever longer) prior to apheresis; 7.Active interstitial lung disease/pneumonitis at the time of ICF signing; 8.Subjects whom the Investigator considers unable to comply with the study protocol or who are otherwise not an appropriate candidate for the study for any reason;

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate after S1904 infusion [Effectiveness] | 3 months
  Independent Review Committee (IRC)-assessed ORR (CR + CRi) at Month 3 post-infusion, as per ALL Response Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, Principal Investigator — Peking University People's Hospital; Hongsheng Zhou, Principal Investigator — Nanfang Hospital, Southern Medical University; Ruidong Zhang, Principal Investigator — Beijing Children's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China